CLINICAL TRIAL: NCT03388203
Title: LC-MS/MS Based 25(OH)D Status in a Large Central European Outpatient Cohort- Gender and Age Specific Differences
Brief Title: LC-MS/MS 25(OH)D Status in a Large Cohort
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Bolzano (Other)
Responsible Party: Principal Investigator, Silvia Giuliani, Department of Clinical Pathology, Azienda Ospedaliera di Bolzano
Other Study IDs: 0055719-BZ
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: 25(OH)D Measurement and 25(OH)D Deficiency
Keywords: 25(OH)D; PTH; mass spectrometry; data mining

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 25(OH)D measurement, PTH measurement — 25(OH)D analyses by LC-MS/MS were performed as part of our routine clinical work with a commercial kit from Recipe (Munich, Germany) ; PTH was measured in lithium-heparin plasma using the PTH STAT assay from Roche Diagnostics (Mannheim, Germany) on a Cobas 8000 auto-analyzer.

SUMMARY:
The present study assessed serum 25(OH)D in a cohort of 74235 outpatients by liquid-chromatography-tandem-mass-spectrometry (LC-MS/MS).

The investigators studied the distribution of serum 25(OH)D concentrations in males and females of different age groups, the prevalence of measurable amounts of 25(OH)D2 and seasonal variability.

DETAILED DESCRIPTION:
Measurements were performed under routine circumstances. Samples were collected in serum tubes with clot-activator. As per routine procedure, samples were centrifuged upon arrival in the lab and stored at 4° C until measurement. 25(OH)D3 and 25(OH)D2 were quantitated separately. Results from subjects <18 years were excluded from the analysis. The study was approved by the local Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* >18 years, outpatients;

Exclusion Criteria:

* <18 years, inpatients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators analyzed retrospectively all serum 25(OH)D results from outpatients ( >18 years ) that were generated between January 1, 2015 and December 31, 2016 at the Central Laboratory of Clinical Pathology at the Bolzano Hospital (Italy). Out of 74,235 samples 3,801 cases were identified where PTH was requested at the same occasion.
Sampling Method: Probability Sample
Enrollment: 74235 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
25(OH)D measurement | 2015-2016
  Describe the 25(OH)D status in South-Tyrol,a region in central Europe, by a rigorously controlled, NIST 972a aligned LC-MS/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: MARKUS HERRMANN, Medicine, Principal Investigator — Clinical Institute for Medical and Chemical Laboratory Diagnostics, Medical University of Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giovannucci E, Liu Y, Rimm EB, Hollis BW, Fuchs CS, Stampfer MJ, Willett WC. Prospective study of predictors of vitamin D status and cancer incidence and mortality in men. J Natl Cancer Inst. 2006 Apr 5;98(7):451-9. doi: 10.1093/jnci/djj101. PMID 16595781
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Yetley EA. Assessing the vitamin D status of the US population. Am J Clin Nutr. 2008 Aug;88(2):558S-564S. doi: 10.1093/ajcn/88.2.558S. PMID 18689402
- [Background] Powe CE, Karumanchi SA, Thadhani R. Vitamin D-binding protein and vitamin D in blacks and whites. N Engl J Med. 2014 Feb 27;370(9):880-1. doi: 10.1056/NEJMc1315850. No abstract available. PMID 24571762
- [Background] Farrell CJ, Martin S, McWhinney B, Straub I, Williams P, Herrmann M. State-of-the-art vitamin D assays: a comparison of automated immunoassays with liquid chromatography-tandem mass spectrometry methods. Clin Chem. 2012 Mar;58(3):531-42. doi: 10.1373/clinchem.2011.172155. Epub 2012 Jan 9. PMID 22230812
- [Background] Farrell C, Soldo J, Williams P, Herrmann M. 25-Hydroxyvitamin D testing: challenging the performance of current automated immunoassays. Clin Chem Lab Med. 2012 Nov;50(11):1953-63. doi: 10.1515/cclm-2012-0522. PMID 23113977
- [Background] Hilger J, Friedel A, Herr R, Rausch T, Roos F, Wahl DA, Pierroz DD, Weber P, Hoffmann K. A systematic review of vitamin D status in populations worldwide. Br J Nutr. 2014 Jan 14;111(1):23-45. doi: 10.1017/S0007114513001840. Epub 2013 Aug 9. PMID 23930771